CLINICAL TRIAL: NCT06525545
Title: Comparison of Clinical and Radiological Results of Patients Undergoing Total Ankle Arthroplasty and Treated With Early Mobilization or With Cast Immobilization
Brief Title: Early MOtion Total Ankle Artroplasty
Acronym: EMOTAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Antonio Mazzotti, Principal Investigator, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMOTAA
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Ankle Osteoarthritis; Ankle - Recurrent Dislocation; Cartilage Disease; Ankle Arthropathy
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Intervention Model Description: interventional randomized case control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilizzazione Precoce (Experimental): early motion of the ankle
  Interventions: Procedure: early mobilizzation of the ankle
- Immobilizzazione Con Stivaletto Gessato (Active Comparator): standard treatment
  Interventions: Procedure: early mobilizzation of the ankle

INTERVENTIONS:
Procedure: early mobilizzation of the ankle — perform flexion-extension exercises of the operated ankle

SUMMARY:
Evaluate the clinical and radiographic results of patients undergoing total ankle arthroplasty and treated in the post-operative period in a randomized manner with early mobilization of the ankle joint or with cast immobilization for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged between 18 and 80).
* Male or female patients;
* Signature of the informed consent for participation in the study;
* Patients prepared and motivated to comply with the scheduled follow-up visits and the completion of the study questionnaires

Exclusion Criteria:

* main diagnosis other than osteoarthritis, history of ankle infection
* need to carry out surgical interventions associated with total prosthesis ankle (e.g., calcaneal osteotomy, knee lowering osteotomy).

first metatarsal bone, supramalleolar osteotomy, etc.)

* intraoperative complications (for example a malleolar fracture) which require a different post-operative protocol
* peripheral vascular disease
* marked osteoporosis of the ankle and foot
* osteonecrosis of the talus
* neurological disorders affecting the lower limb inability to understand study information or respond to questionnaires due to cognitive or linguistic deficits
* patients who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
MOXFQ | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
SF-36 Questionnaire o Short Form-36 Health Survey | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  The 36-Item Short Form Health Survey (SF-36) is a popular questionnaire for measuring the self- erception of quality of life in a given population of interest. Processing the answers of a participant comprises the calculation of 10 scores corresponding to 8 scales measuring several aspects of perceived health and 2 summary components (physical and mental)The scores range from 0 point (best) to 100 (worst).
VAS | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  A Visual Analogue Scale (VAS) is a pain rating scales and ranges from 0 to 10 points
STTA - Sagittal TibioTalar Angle | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  In a lateral weight-bearing radiograph, the saggittal Tibio Talar Angle is the angke between the rantomica axis of the tibia and the he longitudinal axis of the talus, this is determined by drawing a line connecting the midpoints of a line bisecting the talar neck and another line bisecting the talar body
Hindfoot Alignment - Saltzman view mesurament | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  On the saltzman radiologial view is calculated thedistance between the axis of the tibia shaft and the contact point of the heel. Normal values -3 ± 7 mm
Lateral distal tibial angle - LDTA | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  Lateral distal tibia angle (LDTA) is measured between the mid-diaphyseal line of the tibia and the line parallel to the distal tibial plafond. The lateral distal tibial angle has a norm of 89 degrees ± 3 degrees
Anterior distal tibial angle - ADTA | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  The ADTA is formed by the mechanical axis of the tibia and the joint orientation line of the ankle in the sagittal plane and measures 80° ± 3° in the normal lower extremity
Tibio-Talar Angle - TTA | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  The tibiotalar angle is between the anatomic axis of the tibia and the superior articular surface of the talar dome. The mean and standard deviation are: 88.7° ± 5.1°
Center of Rotation of Angulation CORA | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  The CORA is the intersection of the mid-diaphyseal line and the line starting from the middle of the joint and perpendicular to the abnormal ADTA or LDTA. The CORA can be located at the joint line level (usually due to anatomical joint line malalignment or to ankle degeneration) or proximally (usually due to tibial deformities/fractures).
Gamma Angle | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  Gamma angle (γ) is formed by intersection of line drawn through long axis of talar component with line drawn from posterior talar component through middle of talar neck.
T-T ratio (Tibio-talar Ratio) | 3, 6 weeks, 3 - 6 - 9 - 12 - 24 month from the surgery
  Tibiotalar ratio (TT ratio). A talar reference line is drawn parallel to the floor from the posterior talar point (defined as the intersection between the posterosuperior calcaneal cortex and the posterior subtalar articular surface) to the anterior talar point (vertical projection of the most anterior point of the talus onto the talar reference line). Next, the distal tibial axis is the line drawn between the midpoint of the distal tibial shaft measured 5 and 10 cm above the ankle. This divides the talar reference line into anterior and posterior segments. The TT ratio is the ratio of the length of the posterior segment of the talus (AC) to the longitudinal talar length (AB), expressed as a percentage. Normal value, 27% to 42%

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hintermann B, Knupp M, Zwicky L, Barg A. Total ankle replacement for treatment of end-stage osteoarthritis in elderly patients. J Aging Res. 2012;2012:345237. doi: 10.1155/2012/345237. Epub 2012 Jun 5. PMID 22720158
- [Background] Giannini S, Romagnoli M, O'Connor JJ, Catani F, Nogarin L, Magnan B, Malerba F, Massari L, Guelfi M, Milano L, Volpe A, Rebeccato A, Leardini A. Early clinical results of the BOX ankle replacement are satisfactory: a multicenter feasibility study of 158 ankles. J Foot Ankle Surg. 2011 Nov-Dec;50(6):641-7. doi: 10.1053/j.jfas.2011.06.003. Epub 2011 Aug 15. PMID 21840736
- [Background] Mosca M, Caravelli S, Vocale E, Maitan N, Grassi A, Massimi S, Fuiano M, Zaffagnini S. Clinical-radiological outcomes and complications after total ankle replacement through a lateral transfibular approach: a retrospective evaluation at a mid-term follow-up. Int Orthop. 2021 Feb;45(2):437-443. doi: 10.1007/s00264-020-04709-4. Epub 2020 Jul 14. PMID 32666242
- [Background] Onggo JR, Nambiar M, Phan K, Hickey B, Galvin M, Bedi H. Outcome after total ankle arthroplasty with a minimum of five years follow-up: A systematic review and meta-analysis. Foot Ankle Surg. 2020 Jul;26(5):556-563. doi: 10.1016/j.fas.2019.07.006. Epub 2019 Jul 25. PMID 31420116
- [Background] Izzo A, Di Gennaro D, Sgadari A, Coviello A, Marasco D, Balato G, Mariconda M, Bernasconi A. Periprosthetic joint infection in total ankle replacement: which are the current diagnostic criteria? Acta Biomed. 2023 Aug 3;94(4):e2023105. doi: 10.23750/abm.v94i4.14082. PMID 37539613